CLINICAL TRIAL: NCT04386096
Title: Randomized Controlled Trial of Web Based Tools to Improve Medication Continuity in Adolescents With ADHD
Brief Title: Web Based Tools to Improve Medication Continuity in Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020-0236; R34MH112648 (NIH)
Record Dates: First submitted 2020-05-05; First posted 2020-05-13 (Actual); Results first posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-02

CONDITIONS: Attention Deficit Hyperactivity Disorder; Adherence, Medication
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mehealth for ADHD software with medication continuity tools (Experimental)
  Interventions: Other: Mehealth for ADHD software with medication continuity tools
- Mehealth for ADHD software with no medication continuity tools (Active Comparator)
  Interventions: Other: Mehealth for ADHD software with no medication continuity tools

INTERVENTIONS:
Other: Mehealth for ADHD software with medication continuity tools — Medication continuity tools integrated within the mehealth for ADHD software will assess factors influencing medication continuity for each adolescent and recommend tools to address relevant factors. Tools include 1) a system to track outcomes and resolve uncertainty about the need for and/or benefit from medicine, 2) a module to address stigma, 3) a module to help manage side effects, and 4) reminders to take medicine and/or request refills.
  Arms: Mehealth for ADHD software with medication continuity tools
Other: Mehealth for ADHD software with no medication continuity tools — The mehealth for ADHD software has multiple functionalities including 1) online training regarding the American Academy of Pediatrics (AAP) ADHD guidelines; 2) an ADHD workflow wizard that guides pediatricians through the creation of an efficient office workflow to deliver quality ADHD care; 3) online collection of parent- and teacher-report ADHD rating scales for the assessment of ADHD as well as monitoring response to medication treatment; 4) integrated algorithms that automatically score rating scales in real time and provide pediatricians with assessment and treatment reports as well as immediate warnings; 5) an online pediatrician "report card"; and 6) a Plan-Do-Study-Act wizard that allows pediatricians to select a practice behavior to improve based on their report card and guides them through the creation of small tests of change to improve their office systems.
  Arms: Mehealth for ADHD software with no medication continuity tools

SUMMARY:
Medication is an efficacious treatment strategy for adolescents with attention-deficit/hyperactivity disorder (ADHD), however use significantly declines during adolescence when the consequences of ADHD are most severe (e.g. dropping out of school, delinquency, etc.). The Unified Theory of Behavior Change (UTBC) has been proposed as a conceptual model to explain the mechanism underlying ADHD medication adherence and to guide the development of interventions to improve the continuity of treatment. The UTBC is a well-established and empirically tested model that identifies factors that influence an individual's intention to perform a behavior as well as factors that influence whether a behavior is actually carried out. Indeed, the research team's preliminary data support the relevance of pre-intention factors and implementation factors for medication continuity among adolescents with ADHD. Currently, no evidence-based interventions target medication continuity for adolescents with ADHD. The objective of this study is to test a multi-component intervention that systematically identifies and targets aspects of the UTBC model most relevant for each adolescent with poor ADHD medication continuity. The central hypothesis is that the tailored intervention will support ADHD medication continuity. The study will objectively test the central hypothesis by conducting a randomized controlled trial among adolescents with poor medication continuity to test whether the intervention engages the mechanism underlying medication continuity and improves outcomes.

ELIGIBILITY:
Inclusion Criteria:

* First prescribed ADHD medicine more than one year prior to enrollment
* Treated by pediatrician at practice participating in study
* Filled at least one prescription for a stimulant medication in the past year

Exclusion Criteria:

* More than 80% of days covered with medicine over past one year
* Poor understanding level: The participant and parent cannot understand or follow instructions given in the study.
* Do not have reliable access to the internet at their home or another location.
* Parent will not permit their child to access the internet for study related activities
* Are not able or willing to send or receive text messages for study related activities

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mehealth for ADHD Software With Medication Continuity Tools | Mehealth for ADHD Software With no Medication Continuity Tools
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mehealth for ADHD Software With Medication Continuity Tools | Mehealth for ADHD Software With no Medication Continuity Tools | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years]
  Adolescent | 13.17 (1.28) | 13.49 (1.14) | 13.33 (1.20)
  Parent | 37.14 (6.58) | 38.81 (7.07) | 37.98 (6.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Adolescent: Female | 6 | 4 | 10
  Adolescent: Male | 14 | 16 | 30
  Parent: Female | 20 | 20 | 40
  Parent: Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Adolescent: Hispanic or Latino | 2 | 0 | 2
  Adolescent: Not Hispanic or Latino | 17 | 20 | 37
  Adolescent: Unknown or Not Reported | 1 | 0 | 1
  Parent: Hispanic or Latino | 1 | 0 | 1
  Parent: Not Hispanic or Latino | 19 | 20 | 39
  Parent: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Adolescent: American Indian or Alaska Native | 0 | 0 | 0
  Adolescent: Asian | 0 | 0 | 0
  Adolescent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Adolescent: Black or African American | 15 | 17 | 32
  Adolescent: White | 2 | 2 | 4
  Adolescent: More than one race | 3 | 1 | 4
  Adolescent: Unknown or Not Reported | 0 | 0 | 0
  Parent: American Indian or Alaska Native | 0 | 0 | 0
  Parent: Asian | 0 | 0 | 0
  Parent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Parent: Black or African American | 15 | 14 | 29
  Parent: White | 4 | 2 | 6
  Parent: More than one race | 1 | 3 | 4
  Parent: Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Days Covered With Medicine
Description: This will be calculated based pharmacy dispensing records
Time Frame: An average of 4 months
Measure: Median (Full Range); unit: proportion of days covered with medicine
Arm/Group | Mehealth for ADHD Software With Medication Continuity Tools | Mehealth for ADHD Software With no Medication Continuity Tools
Number analyzed (Participants) | 20 | 20
proportion of days covered with medicine | 0.24 [0 to 0.97] | 0 [0 to 0.63]
Statistical Analysis 1: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Fidelity to Intended Use of Intervention Components
Description: Proportion of intervention components completed relative to the components that were recommended by the portal based on adolescent/parent responses to the assessment battery.
Time Frame: An average of 4 months
Population: Data were only collected for the "Mehealth for ADHD software with medication continuity tools" group
Measure: Mean (Full Range); unit: Proportion of intervention components
Arm/Group | Mehealth for ADHD Software With Medication Continuity Tools | Mehealth for ADHD Software With no Medication Continuity Tools
Number analyzed (Participants) | 20 | 0
Proportion of intervention components | 0.07 [0.0 to 0.60] |

3. Secondary Outcome: Change in Pre-intention Factors of Unified Theory of Behavior Change
Description: Adolescent and parent self-report on a 1-5 or 1-7-point scale, depending on the item. Items were re-scaled to a 1 (signifying less belief) to 5 (signifying stronger belief) scale. Individual items measure specific attitudes, subjective norms, and perceived behavioral control. Items were coded so that higher scores aligned with increased perceived advantages of performing the behavior and behavioral control around taking ADHD medicine. We calculated the average score of the total items (Adolescent report = 19 items; Parent report = 17 items). Range of change score is (-4) to (+4).
Time Frame: At baseline and approximately 4 months later
Population: Missing data for 2 participants in the "Mehealth for ADHD software with no medication continuity tools" group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mehealth for ADHD Software With Medication Continuity Tools | Mehealth for ADHD Software With no Medication Continuity Tools
Number analyzed (Participants) | 20 | 18
score on a scale
  Adolescent | -0.08 (0.55) | 0.14 (0.72)
  Parent | -0.24 (0.46) | -0.18 (0.54)
Statistical Analysis 1: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Adolescent Pre-Intention Factors; Test type: Superiority; p = 0.30, t-test, 2 sided
Statistical Analysis 2: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Parent Pre-Intention Factors; Test type: Superiority; p = 0.71, t-test, 2 sided

4. Secondary Outcome: Change in Intention to Take/Give ADHD Medicine Regularly
Description: Adolescent and parent self-report on a 1-7-point scale. Items were re-scaled to a 1 (signifying less intention) to 5 (signifying stronger intention) scale. Items were coded so that higher scores aligned with stronger intention to take ADHD medicine every school day, weekend day, and during school vacations. We calculated the average score of the 3 items. Range of change score is (-4) to (+4).
Time Frame: At baseline and approximately 4 months later
Population: Missing data for 2 participants in the "Mehealth for ADHD software with no medication continuity tools" group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mehealth for ADHD Software With Medication Continuity Tools | Mehealth for ADHD Software With no Medication Continuity Tools
Number analyzed (Participants) | 20 | 18
score on a scale
  Adolescent | -0.51 (1.4) | -0.01 (1.43)
  Parent | 0.03 (1.19) | -0.42 (0.86)
Statistical Analysis 1: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Adolescent Intention to take/give ADHD medicine regularly; Test type: Superiority; p = 0.29, t-test, 2 sided
Statistical Analysis 2: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Parent Intention to take/give ADHD medicine regularly; Test type: Superiority; p = 0.19, t-test, 2 sided

5. Secondary Outcome: Change in Adolescent-report of Medication Barriers
Description: Adolescent self-report on Adolescent Medication Barriers Scale using a 1-5-point Likert Scale. 1 indicates strong agreement and 5 indicates strong disagreement, with higher scores indicating less barriers. Items were coded so that higher scores aligned with increased organizational skills, salience of behavior, and routine around taking ADHD medicine. We calculated the average score of the 8 items. Range of change score is (-4) to (+4).
Time Frame: At baseline and approximately 4 months later
Population: Missing data for 2 participants in the "Mehealth for ADHD software with no medication continuity tools" group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mehealth for ADHD Software With Medication Continuity Tools | Mehealth for ADHD Software With no Medication Continuity Tools
Number analyzed (Participants) | 20 | 18
score on a scale | 0.08 (0.76) | 0.19 (0.8)
Statistical Analysis 1: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Test type: Superiority; p = 0.64, t-test, 2 sided

6. Secondary Outcome: Change in Parent-report of Medication Barriers
Description: Parent self-report on Parent Medication Barriers Scale using a 1-5-point Likert Scale. 1 indicates strong agreement and 5 indicates strong disagreement, with higher scores indicating less barriers. Items were coded so that higher scores aligned with increased adolescent organizational skills, salience of behavior, and routine around taking ADHD medicine. We calculated the average score of the 9 items. Range of change score is (-4) to (+4).
Time Frame: At baseline and approximately 4 months later
Population: Missing data for 2 participants in the "Mehealth for ADHD software with no medication continuity tools" group. One participant in the "Mehealth for ADHD software with no medication continuity tools" group did not respond to one survey item.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mehealth for ADHD Software With Medication Continuity Tools | Mehealth for ADHD Software With no Medication Continuity Tools
Number analyzed (Participants) | 20 | 18
score on a scale | -0.11 (0.5) | -0.07 (0.61)
Statistical Analysis 1: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Test type: Superiority; p = 0.81, t-test, 2 sided

7. Secondary Outcome: Change in Medication Diversion
Description: Adolescent self-report of the number of occasions of giving away, trading, or selling ADHD medicine to someone for whom it was not prescribed.
Time Frame: At baseline and approximately 4 months later
Population: Missing data for 2 participants in the "Mehealth for ADHD software with no medication continuity tools" group
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Mehealth for ADHD Software With Medication Continuity Tools | Mehealth for ADHD Software With no Medication Continuity Tools
Number analyzed (Participants) | 20 | 18
Events | 0 (0) | 0 (0)

8. Secondary Outcome: Change in Decision Making Involvement Scale
Description: Adolescent and Parent self-report. The scale contains the following subscales: "Child Seek" (e.g. child asks for an opinion or information from the parent), "Child Express" (e.g. child expresses an opinion or information to the parent), "Parent Seek" (e.g. parent asks for an opinion or information from child), "Parent Express" (e.g. parent expresses advice, an opinion, or information to the child), and "Joint/Options" (e.g. negotiation and brainstorming between child and parent). Each subscale produces a score which ranges from 1 to 4 with higher scores indicating more of that behavior.
Time Frame: At baseline and approximately 4 months later
Population: Missing data for 2 participants in the "Mehealth for ADHD software with no medication continuity tools" group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mehealth for ADHD Software With Medication Continuity Tools | Mehealth for ADHD Software With no Medication Continuity Tools
Number analyzed (Participants) | 20 | 18
score on a scale
  Adolescent: Child Seek | -0.02 (1.02) | -0.02 (1.20)
  Adolescent: Child Express | 0 (1.12) | 0.24 (1.12)
  Adolescent: Parent Seek | 0.16 (0.82) | 0.10 (1.16)
  Adolescent: Parent Express | 0.13 (0.90) | 0.10 (1.04)
  Adolescent: Joint/Options | 0.02 (0.91) | 0.27 (1.01)
  Parent: Child Seek | -0.05 (0.96) | -0.07 (0.85)
  Parent: Child Express | -0.07 (1.02) | -0.15 (0.81)
  Parent: Parent Seek | -0.10 (0.66) | -0.22 (0.79)
  Parent: Parent Express | -0.11 (0.82) | -0.11 (0.71)
  Parent: Joint/Options | -0.05 (0.88) | -0.04 (0.80)
Statistical Analysis 1: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Adolescent: Child Seek; Test type: Superiority; p = 0.10, t-test, 2 sided
Statistical Analysis 2: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Adolescent: Child Express; Test type: Superiority; p = 0.51, t-test, 2 sided
Statistical Analysis 3: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Adolescent: Parent Seek; Test type: Superiority; p = 0.84, t-test, 2 sided
Statistical Analysis 4: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Adolescent: Parent Express; Test type: Superiority; p = 0.93, t-test, 2 sided
Statistical Analysis 5: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Adolescent: Joint/Options; Test type: Superiority; p = 0.43, t-test, 2 sided
Statistical Analysis 6: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Parent: Child Seek; Test type: Superiority; p = 0.94, t-test, 2 sided
Statistical Analysis 7: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Parent: Child Express; Test type: Superiority; p = 0.79, t-test, 2 sided
Statistical Analysis 8: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Parent: Parent Seek; Test type: Superiority; p = 0.61, t-test, 2 sided
Statistical Analysis 9: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Parent: Parent Express; Test type: Superiority; p = 0.10, t-test, 2 sided
Statistical Analysis 10: Comparison: Mehealth for ADHD Software With Medication Continuity Tools vs Mehealth for ADHD Software With no Medication Continuity Tools; Change in Parent: Joint/Options; Test type: Superiority; p = 0.98, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Mehealth for ADHD Software With Medication Continuity Tools | Mehealth for ADHD Software With no Medication Continuity Tools
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT04386096/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT04386096/SAP_001.pdf
  • Informed Consent Form (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT04386096/ICF_002.pdf